CLINICAL TRIAL: NCT07261644
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of 608 in Adult Subjects With Active Ankylosing Spondylitis (AS)
Brief Title: A Study to Evaluate the Efficacy and Safety of 608 in Adult Subjects With Active Ankylosing Spondylitis(AS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-608-AS-III-01
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 608 Dose (Experimental): 608 subcutaneous (SC) injection.
  Interventions: Drug: 608 dose
- Placebo (Placebo Comparator): Placebo subcutaneous (SC) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 608 dose — 608 subcutaneous (SC) injection.
  Arms: 608 Dose
Drug: Placebo — Placebo subcutaneous (SC) injection.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of 608 in patients with AS.

DETAILED DESCRIPTION:
The purpose of this trial is to demonstrate the clinical efficacy at week 16; and to demonstrate safety and tolerability of 608 compared to placebo in patients with ankylosing spondylitis at week 16 and long term safety up to Week 60.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the protocol requirements, participate and sign the informed consent form (ICF) voluntarily;
2. At least 18 years of age at the time of signing the ICF, with no gender restrictions;
3. Meet the 1984 modified New York criteria for ankylosing spondylitis (AS);
4. Have inadequate response to non-steroidal anti-inflammatory drugs (NSAIDs) or have contraindications/intolerance to NSAIDs treatment;
5. Willing to practice contraception and have no plans for pregnancy, sperm donation, or egg donation from the screening period until at least 6 months after the last dose.

Exclusion Criteria:

1. Patients with other uncontrolled active inflammatory diseases.
2. Clinical laboratory tests and other tests that reveal abnormalities with clinical significance
3. Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
4. History of cancer.
5. Known or suspected history of immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 40 Response. | Week 16.
  Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a NRS; 2. Patient's assessment of back pain, measured on a NRS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by NRS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by NRS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant). ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the NRS signifies higher severity.

SECONDARY OUTCOMES:
The Percentage of Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 20 Response. | Week 16.
  Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a NRS; 2. Patient's assessment of back pain, measured on a NRS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by NRS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by NRS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant). ASAS 20 response is defined as an improvement of ≥20% and ≥1 unit on a scale of 10 in at least three of the four main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain. A higher score on the NRS signifies higher severity.

OTHER OUTCOMES:
608 Concentration in Serum. | Up to 60 Weeks.
  The concentration of 608 in Serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No